CLINICAL TRIAL: NCT01734408
Title: A Booster Dose of Inactivated Vaccine (Vero Cell) Against EV71 in Chinese Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Collaborators: Bejing Vigoo Biological Co., LTD (Industry)
Responsible Party: Principal Investigator, Fengcai Zhu, vice director, Jiangsu Province Centers for Disease Control and Prevention
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: JSVCT005b
Record Dates: First submitted 2012-11-22; First posted 2012-11-27 (Estimated); Last update posted 2013-10-23 (Estimated); Status verified 2013-10

CONDITIONS: EV71-associated Disease
Keywords: immunogenicity; safety; inactivated EV71 vaccine
MeSH Terms: interventions — Aluminum Hydroxide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- alum-adjuvant 160U /0.5ml EV71 vaccine (Experimental): A booster dose of alum-adjuvant 160U /0.5ml EV71 vaccine in 160 children whom had received two doses of alum-adjuvant 160U/0.5ml EV71 vaccines one year before.
  Interventions: Biological: alum-adjuvant 160U /0.5ml
- placebo A (Placebo Comparator): A 0/0.5ml placebo in 80 children whom had received two doses of alum-adjuvant 160U/0.5ml EV71 vaccines one year before.
  Interventions: Biological: 0/0.5ml placebo
- alum-adjuvant 320U /0.5ml EV71 vaccine (Experimental): A booster dose of alum-adjuvant 320U /0.5ml EV71 vaccine in 160 children whom had received two doses of alum-adjuvant 320U/0.5ml EV71 vaccines one year before.
  Interventions: Biological: alum-adjuvant 320U /0.5ml
- placebo B (Placebo Comparator): A 0/0.5ml placebo in 80 children whom had received two doses of alum-adjuvant 320U/0.5ml EV71 vaccines one year before.
  Interventions: Biological: 0/0.5ml placebo
- alum-adjuvant 640U /0.5ml EV71 vaccine (Experimental): A booster dose of alum-adjuvant 640U /0.5ml EV71 vaccine in 160 children whom had received two doses of alum-adjuvant 640U/0.5ml EV71 vaccines one year before.
  Interventions: Biological: alum-adjuvant 640U /0.5ml
- placebo C (Placebo Comparator): A 0/0.5ml placebo in 80 children whom had received two doses of alum-adjuvant 640U/0.5ml EV71 vaccines one year before.
  Interventions: Biological: 0/0.5ml placebo
- adjuvant-free 640U /0.5ml EV71 vaccine (Experimental): A booster dose of adjuvant-free 640U /0.5ml EV71 vaccine in 160 children whom had received two doses of adjuvant-free 640U/0.5ml EV71 vaccines one year before.
  Interventions: Biological: adjuvant-free 640U /0.5ml
- placebo D (Placebo Comparator): A 0/0.5ml placebo in 80 children whom had received two doses of adjuvant-free 640U/0.5ml EV71 vaccines one year before.
  Interventions: Biological: 0/0.5ml placebo

INTERVENTIONS:
Biological: alum-adjuvant 160U /0.5ml — inactivated vaccine (vero cell) alum-adjuvant 160U /0.5ml EV71 vaccine
  Arms: alum-adjuvant 160U /0.5ml EV71 vaccine
Biological: alum-adjuvant 320U /0.5ml — inactivated vaccine (vero cell) alum-adjuvant 320U /0.5ml EV71 vaccine
  Arms: alum-adjuvant 320U /0.5ml EV71 vaccine
Biological: alum-adjuvant 640U /0.5ml — inactivated vaccine (vero cell) alum-adjuvant 640U /0.5ml EV71 vaccine
  Arms: alum-adjuvant 640U /0.5ml EV71 vaccine
Biological: adjuvant-free 640U /0.5ml — inactivated vaccine (vero cell) adjuvant-free 640U /0.5ml EV71 vaccine
  Arms: adjuvant-free 640U /0.5ml EV71 vaccine
Biological: 0/0.5ml placebo — 0/0.5ml placebo
  Arms: placebo A; placebo B; placebo C; placebo D

SUMMARY:
Hand, foot, and mouth disease (HFMD) is a common viral illness in infants and children caused by viruses that belong to the enterovirus genus of the picornavirus family. Although most HFMD cases do not result in serious complications, outbreaks of HFMD caused by enterovirus 71 (EV71) can present with a high rate of neurological complications, including meningoencephalitis, pulmonary complications, and can even cause infant death. HFMD caused by EV71 has become a major emerging infectious disease in Asia and the highly pathogenic potential of EV71 clearly requires the attention of world medical community.

The phase II study of inactivated vaccine (vero cell) against EV71 has completed last month in Jiangsu Province in China. The data from the phase II study suggested that the inactivated EV71 vaccine had a clinically acceptable safety and good immunogenicity for healthy Chinese children and infants. But the antibody titer against EV71 was found decreased significantly at month 8 compared to that at day 56. Considering the similar dynamic trend had also been found in the antibody against poliovirus induced by polio vaccines, and whose immunization schedule contains a booster dose administrated at 1 to 1.5 year after the first 3 doses of fundamental immunity. In order to find a better immunization schedule for children, the investigators decided to perform this booster immunity trial among these children who had received two doses of EV71 vaccines (around one year after the fundamental immunity). The investigators do the recruitment among these children who had participated in the previous phase II trial and received EV71 vaccines, and randomize them in a ratio of 2:1 to receive either a booster dose of EV71 vaccines or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Had participated in the previous phase II trial and received at least 1 dose of EV71 vaccine.
* Healthy children as established by medical history and clinical examination
* The subjects' guardians are able to understand and sign the informed consent
* Subjects who can and will comply with the requirements of the protocol
* Subjects with temperature <=37.0°C on axillary setting

Exclusion Criteria:

* Had participated in the previous phase II trial and received placebo.
* Subject who has a medical history of EV71-associated disease with specific laboratory evidence
* <= 37 weeks gestation
* Subjects with a birth weight <2.5 kg
* Subject that has a medical history of any of the following: allergic history, or allergic to any ingredient of vaccine
* Family history of seizures or progressive neurological disease
* Family history of congenital or hereditary immunodeficiency
* Severe malnutrition or dysgenopathy
* Major congenital defects or serious chronic illness, including perinatal brain damage
* Autoimmune disease
* Bleeding disorder diagnosed by a doctor or significant bruising or bleeding difficulties with IM injections or blood draws
* Any acute infections in last 7 days
* Any prior administration of immunodepressant or corticosteroids in last 6month
* Any prior administration of blood products in last 3 month
* Any prior administration of other research medicines in last 1 month
* Any prior administration of attenuated live vaccine in last 14 days
* Any prior administration of subunit or inactivated vaccines in last 7 days, such as pneumococcal vaccine
* Under the anti-TB prevention or therapy
* Any condition that in the opinion of the investigator, may interfere with the evaluation of study objectives

Ages: 21 Months to 51 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 773 (Actual)
Dates: Start 2012-11; Primary Completion 2013-01 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Geometric mean titer (GMT) of anti-EV71 antibodies | 28 days after vaccination
  GMT of anti-EV71 antibodies in serum 28 days after booster dose injection

SECONDARY OUTCOMES:
Safety of EV71 vaccine in healthy children | 28 days after vaccination
  Frequency of systemic and local adverse reactions in healthy children following 28 days after the boosting dose of EV71 vaccine
Geometric mean fold increase (GMFI) of anti-EV71 antibodies | 28 days after vaccination
  GMFI of anti-EV71 antibodies in serum 28 days after vaccination
Seroconversion of anti-EV71 antibodies | 28 days after vaccination
  Seroconversion of anti-EV71 antibodies in serum 28 days after vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Provincial Center for Diseases Control and Prevention, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Shenyu W, Jingxin L, Zhenglun L, Xiuling L, Qunying M, Fanyue M, Hua W, Yuntao Z, Fan G, Qinghua C, Yuemei H, Xin Y, Huijie G, Fengcai Z. A booster dose of an inactivated enterovirus 71 vaccine in chinese young children: a randomized, double-blind, placebo-controlled clinical trial. J Infect Dis. 2014 Oct 1;210(7):1073-82. doi: 10.1093/infdis/jiu113. Epub 2014 Mar 12. PMID 24625805